CLINICAL TRIAL: NCT04737200
Title: The Impact of Overnight Nutrition Support on Sleep and Circadian Rhythm Disruption in the ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hassan Dashti, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020P003989
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Feeding Patterns; Sleep; Glucose Intolerance
Keywords: Enteral Nutrition; Chrononutrition; Intensive Care Unit; Chronobiology; Nutrition Support; Sleep
MeSH Terms: conditions — Feeding Behavior; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nighttime cycled enteral feeds first (Experimental): Patients will start nighttime cycled enteral feeds first for 12 hours. Following a 24-hour washout period, patients will then start daytime cycled enteral feeds for 12 hours.
  Interventions: Dietary Supplement: Time-of-day of enteral nutrition provision (nighttime first)
- Daytime cycled enteral feeds first (Experimental): Patients will start daytime cycled enteral feeds first for 12 hours. Following a 24-hour washout period, patients will then start nighttime cycled enteral feeds for 12 hours.
  Interventions: Dietary Supplement: Time-of-day of enteral nutrition provision (daytime first)

INTERVENTIONS:
Dietary Supplement: Time-of-day of enteral nutrition provision (daytime first) — Enteral nutrition (tube feeds) will be provided during the daytime followed by nighttime.
  Arms: Daytime cycled enteral feeds first
Dietary Supplement: Time-of-day of enteral nutrition provision (nighttime first) — Enteral nutrition (tube feeds) will be provided during the nighttime followed by daytime.
  Arms: Nighttime cycled enteral feeds first

SUMMARY:
The purpose of this study is to determine whether modifying the timing of nutrition support from overnight to daytime enhances sleep quality, preserves circadian rhythms, and improves overall inflammation and cardiometabolic profiles in postoperative patients in the cardiac surgical ICU on enteral nutrition.

DETAILED DESCRIPTION:
Intensive care unit (ICU) environments do not support sleep or preserve circadian rhythms of postoperative critically ill patients. Among the contributing factors is the common practice of administering nutrition support through feeding tubes overnight. The overall objective of the study is to examine a novel dimension of clinical nutrition by determining whether enhancing sleep quality and preserving robust circadian rhythms through daytime instead of overnight feeds will attenuate inflammation and improve cardiometabolic profiles of postoperative cardiac ICU patients on nutrition support. The investigators hypothesize that overnight nutrition support results in fragmented sleep and blunted circadian rhythms and thus represent a modifiable mechanism exacerbating inflammation and cardiometabolic derangements in postoperative cardiac patients. Results of this study will help in the development of evidence-based, cost-efficient, and effective enteral nutrition timing countermeasures against fragmented sleep, disrupted circadian rhythms, inflammation and cardiometabolic derangements and potentially modify the current widespread practice of overnight nutrition likely affecting 250,000 hospital admissions annually in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or non-pregnant female volunteers (age 18+)
* Scheduled for a cardiac surgical procedure with planned post-operative admission to the ICU for >48 hours
* Able and willing to give consent and comply with study procedures

Exclusion Criteria:

* Blind, deaf or unable to speak English
* Women who are pregnant or nursing
* Contraindications to safe use enteral nutrition, including gastrointestinal obstruction
* Personal history of intestinal malabsorption, gallbladder disease or pancreatitis
* Dietary restrictions precluding enteral feeds
* Renal and liver failure requiring dialysis or Child-Pugh score > 7
* Severe deficit due to structural or anoxic brain damage
* With skin condition that precludes wearing sensors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Sleep fragmentation | Approximately 12 hours. Estimated from nighttime sleep following daytime cycled enteral feeds and during nighttime cycled enteral feeds.
  Sleep fragmentation is defined as the number of shifts from deeper (N2, N3, REM) to lighter (W or N1) sleep stages by hours of sleep. Sleep fragmentation will be assessed objectively through EEG measures.
Circadian rhythms amplitude | Estimated from data collected 12 hours prior to and the 12 hours during daytime cycled and nighttime cycled enteral feeds.
  Amplitude is defined as peak-to-nadir difference in rhythms estimated from body temperature and actigraphy.

SECONDARY OUTCOMES:
Sleep arousals | Approximately 12 hours. Estimated from nighttime sleep following daytime cycled enteral feeds and during nighttime cycled enteral feeds.
  Sleep arousals is defined as n shifts from N1, N2, N3, REM to wake divided by hours of sleep. Sleep arousals will be assessed objectively through EEG measures.
Total sleep time | Approximately 12 hours. Estimated from nighttime sleep following daytime cycled enteral feeds and during nighttime cycled enteral feeds.
  Measure of sleep duration and assessed objectively through EEG measures.
Duration of sleep stages | Approximately 12 hours. Estimated from nighttime sleep following daytime cycled enteral feeds and during nighttime cycled enteral feeds.
  Duration of the following sleep stages will be estimated: N1, N2, N3, REM sleep. Sleep stages will be assessed objectively through EEG measures.
Sleep midpoint | Approximately 12 hours. Estimated from nighttime sleep following daytime cycled enteral feeds and during nighttime cycled enteral feeds.
  Sleep midpoint is defined as the midpoint between start and end of sleep episode. Sleep midpoint will be determined objectively from EEG measures.
Acrophase | Estimated from data collected 12 hours prior to and the 12 hours during daytime cycled and nighttime cycled enteral feeds.
  Acrophase is defined as the time of peak activity.
Midpoint of least-active 5h timing | Estimated from data collected 12 hours prior to and the 12 hours during daytime cycled and nighttime cycled enteral feeds.
  Measure of sleep timing as determined from actigraphy.
Midpoint of most-active 10h timing | Estimated from data collected 12 hours prior to and the 12 hours during daytime cycled and nighttime cycled enteral feeds.
  Measure of sleep timing as determined from actigraphy.
Inactivity duration | Estimated from data collected 12 hours prior to and the 12 hours during daytime cycled and nighttime cycled enteral feeds.
  Duration of inactivity outside of sleep episode as determined from actigraphy.
12 hours average systolic and diastolic blood pressure | Estimated from data collected 12 hours prior to and the 12 hours during daytime cycled and nighttime cycled enteral feeds.
  Continuously measured using ECG. Systolic and diastolic blood pressure will be averaged during each 12-hour cycled feed.
12 hours average glucose | Estimated from data collected 12 hours prior to and the 12 hours during daytime cycled and nighttime cycled enteral feeds.
  Continuously measured using continuous glucose sensors. Blood glucose will be averaged during each 12-hour cycled feed.
C-reactive protein | Blood draw scheduled at 8 am and 8 pm on days on daytime cycled and nighttime cycled enteral feeds.
  The inflammatory biomarker C-reactive protein will be measured from serum.
Interleukin-6 | Blood draw scheduled at 8 am and 8 pm on days on daytime cycled and nighttime cycled enteral feeds.
  The inflammatory biomarker Interleukin-6 will be measured from serum.
Tumor necrosis factor α | Blood draw scheduled at 8 am and 8 pm on days on daytime cycled and nighttime cycled enteral feeds.
  The inflammatory biomarker Tumor necrosis factor α will be measured from serum.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan S Dashti, Ph.D., R.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dashti HS, Wang YM, Knauert MP. Feeding critically ill patients at the right time of day. Crit Care. 2024 Jun 24;28(1):206. doi: 10.1186/s13054-024-04994-0. No abstract available. PMID 38915028